CLINICAL TRIAL: NCT02839486
Title: Vancomycin and Cefoxitin Levels During Pediatric Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Vancomycin and Cefoxitin During Pediatric Cardiopulmonary Bypass
Acronym: VANCOCEF
Status: Completed | Type: Observational
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Zaccaria Ricci, Medical Doctor, Bambino Gesù Hospital and Research Institute
Other Study IDs: vanco and cefoxitin during CPB
Record Dates: First submitted 2016-07-10; First posted 2016-07-21 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Congenital Heart Disease
Keywords: antibiotic prophylaxis; pharmacokinetics; cardiopulmonary bypass
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- vancomycin and cefoxitin pharmacokinetics: This is surgical prophylaxis and cefoxitin/vancomycin have to be administered to each patient of the study, before surgery
  Interventions: Other: vancomycin pharmacokinetics; Other: cefoxitin pharmacokinetics

INTERVENTIONS:
Other: vancomycin pharmacokinetics — vancomycin serial plasmatic and ultrafiltrate samples in order to assess plasmatic and ultrafiltrate drug concentrations
Other: cefoxitin pharmacokinetics — cefoxitin serial plasmatic and ultrafiltrate samples in order to assess plasmatic and ultrafiltrate drug concentrations

SUMMARY:
The aim of this study will be to evaluate vancomycin and cefoxitin blood levels during elective cardiopulmonary bypass (CPB) surgery in four pre-determined pediatric strata: neonates, infants, children weighting less than 40 kg and children weighting more than 40 kg.

DETAILED DESCRIPTION:
Few data are available in current literature about pharmacokinetics (PK) of antibiotics administered as surgical prophylaxis to children scheduled for cardiac surgery with CPB. In particular, vancomycin PK during CPB has been studied only in small case series, whereas no specific study has been conducted, so far, in the specific setting of children receiving cefoxitin during CPB.

CPB affects patients' volemia and drugs PK is eventually altered. On the other side during and after surgery for heart defects, many risk factors may decrease renal and hepatic clearance, including altered renal perfusion, use of vasoactive agents, and use of concomitant nephrotoxic medications.

Primary Objective of the study will be:

• To study the pharmacokinetic profile of vancomycin and cefoxitin administered, as antibiotic prophylaxis to children undergoing elective CPB.

Secondary Objectives will be:

* To evaluate if a significant difference in blood levels will occur in the four predetermined patients' categories.
* To evaluate the role of hemodilution during CPB on studied antibiotics' serum concentration
* To verify the incidence of post-operative infections in the studied population with particular attention to sensitive bacteria
* To evaluate the impact of ultrafiltration in studied antibiotics' clearance
* To evaluate safety of the administered antibiotics This is a prospective monocentric, open label, not controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Elective cardiac surgery schedule with the planned application of CPB
2. Parents of neonates, or their legal representative, able to consent and comply with protocol requirements.

Exclusion Criteria:

1. Urgent or emergent surgery
2. Antibiotic therapy (any) administered before surgery
3. Patients receiving, before surgery, any other ofr of extracorporeal treatment (i.e extracorporeal membrane oxygenation, continuous renal replacement therapy)
4. Previous renal or hepatic dysfunction requiring need for antibiotic posology modification.
5. Surgery requiring antibiotic prophylaxis with different drug combinations (i.e vancomycin and gentamycin)
6. extremely low birth weight neonates.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing cardiac surgery requiring cardiopulmonary bypass and antibiotic prophylaxis with vancomycin and cefoxitin
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
vancomycin and cefoxitin concentration change in serial plasmatic samples | samples will be withdrawn: at skin incision, 15 minutes after CPB start (CPB1), at the end of CPB (CPB2), at end of surgery.
  a 4-points pharmacokinetic curve per each antibiotic will be generated by serial average plasmatic vancomycin and cefoxitin concentration assessments.

SECONDARY OUTCOMES:
differences between pre-determined subgroups (neonates, infants, children weighting less than 40 kg and children weighting more than 40 kg) in plasmatic vancomycin and cefoxitin levels change at each time point | samples will be withdrawn: at skin incision, 15 minutes after CPB start (CPB1), at the end of CPB (CPB2).
vancomycin and cefoxitin clearance by ultrafiltration | Ultrafiltrate sample will be withdrawn at the end of CPB (UF1)
  The clearance of vancomycin and cefoxitin in the ultrafiltrate (UF) will be evaluated. Antibiotics' sieving coefficient (SC) will be calculated from antibiotics concentrations at the following time points: UF1/[(CPB1+CPB2)/2]. Antibiotics clearance will be calculated as SC*UF rate (ml/min)

CONTACTS AND LOCATIONS:
Overall Officials: zaccaria ricci, MD, Principal Investigator — Bambino Gesù Hospital
Locations (1):
- Terapia Intenisva Cardiochirurgica, Roma, Italy

IPD SHARING:
Plan to Share IPD: No